CLINICAL TRIAL: NCT07328113
Title: Association Between Interleukin-6 and Thyroid Hormone Dysfunction in Patients With Chronic Kidney Disease Undergoing Hemodialysis
Brief Title: Interleukin-6 and Thyroid Dysfunction in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Universitas Airlangga Hospital, Surabaya (Unknown)
Responsible Party: Sponsor
Other Study IDs: 175/KEP/2023
Record Dates: First submitted 2025-11-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease on Hemodialysis; Thyroid Gland Disease
Keywords: Interleukin-6; Thyroid Function; Chronic Kidney Disease; Hemodialysis
MeSH Terms: conditions — Thyroid Diseases; Renal Insufficiency, Chronic | interventions — Thyroid Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thyroid hormone — Sampling was carried out using a consecutive sampling method, in which every patient who met the study criteria was included as a sample until the predetermined sample size was achieved. Patients who had been confirmed to meet the inclusion and exclusion criteria underwent blood collection of 10 mL (serum or plasma) prior to hemodialysis for the examination of complete blood count, BUN, creatinine, albumin, fasting blood glucose, IL-6, FT4, T3, FT3, T4, and TSH.
  The IL-6 level was measured using the Automatic Immunoassay Fluorescence method with the Automatic Fluorescence Immunoassay Analyzer Vazyme QD-S2000. Thyroid function tests (FT4, T3, T4, FT3, and TSH) were performed using the Enzyme-Linked Immunosorbent Assay (ELISA) method with Autobio Immunoassay reagents on the Autobio A1000 analyzer.
  Other Names: Interleukin-6

SUMMARY:
Chronic kidney disease (CKD) is often associated with multiorgan complications, including thyroid hormone dysfunction. Interleukin-6 (IL-6), a pro-inflammatory cytokine, has been proposed as a marker of inflammation that may contribute to these alterations. The main question it aims to answer is:

Is there an association between interleukin-6 and thyroid hormone dysfunction in patients with chronic kidney disease (CKD) Blood samples will be collected and analyzed from 65 patients who have undergone hemodialysis for at least 3 months.

DETAILED DESCRIPTION:
This cross-sectional observational study involves patients with CKD undergoing hemodialysis at Airlangga University Hospital. Data were collected based on their medical record and Blood test for IL-6. Linear regression analysis assessed the relationship between IL-6 levels and thyroid function parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 Years Old and above
* Patients with ESRD who have undergone hemodialysis for ≥ 3 months and are in stable condition.
* Patients are able to communicate and respond to questions appropriately
* Patients are willing to participate in the study.

Exclusion Criteria:

* ESRD patients undergoing hemodialysis who have been diagnosed with underlying thyroid disorders or thyroid malignancy.
* Patients with a history of thyroid surgery or any intervention involving the thyroid gland.
* Patients with a family history of thyroid disorders.
* Patients taking medications that affect thyroid function or using antioxidant drugs.
* Patients with infection or sepsis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population consists of all ESRD patients aged ≥ 21 years who undergo examinations at the Dialysis Unit of Universitas Airlangga Hospital, Surabaya. The accessible population includes all ESRD patients aged ≥ 21 years who undergo examinations at the Dialysis Unit of Universitas Airlangga Hospital, Surabaya, during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation between serum Interleukin-6 (IL-6) concentration and serum Thyroid-Stimulating Hormone (TSH) levels | At baseline, during routine hemodialysis visit (prior to any study-specific intervention)
  Serum IL-6 (pg/mL) and TSH (µIU/mL) will be measured using standardized hospital laboratory immunoassay analyzers. The outcome is the correlation coefficient (Spearman r) between IL-6 and TSH.

SECONDARY OUTCOMES:
Correlation between serum IL-6 concentration and serum Total Triiodothyronine (T3) levels | At baseline, during routine hemodialysis visit (prior to any study-specific intervention)
  Both IL-6 (pg/mL) and T3 (ng/dL) will be measured using immunoassay. The outcome is the Spearman correlation coefficient.
Correlation between serum IL-6 concentration and serum Total Thyroxine (T4) levels | At baseline, during routine hemodialysis visit (prior to any study-specific intervention)
  IL-6 (pg/mL) and total T4 (µg/dL) will be quantified using immunoassay. Outcome is the correlation coefficient (Spearman r).
Correlation between serum IL-6 concentration and Free Triiodothyronine (fT3) levels | At baseline, during routine hemodialysis visit (prior to any study-specific intervention)
  IL-6 (pg/mL) and free T3 (pg/mL) measured using immunoassay analyzer. Outcome is Spearman correlation coefficient.
Correlation between serum IL-6 concentration and Free Thyroxine (fT4) levels | At baseline, during routine hemodialysis visit (prior to any study-specific intervention)
  IL-6 (pg/mL) and fT4 (ng/dL) measured using immunoassay. Outcome is Spearman correlation coefficient (spearman r).

CONTACTS AND LOCATIONS:
Overall Officials: Sony Wibisono Mudjanarko, dr., Sp.PD, K-EMD, PhD, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Airlangga University Hospital, Surabaya, East Java, Indonesia